CLINICAL TRIAL: NCT01182883
Title: A Phase I Study of IMC-A12 (Anti-Insulin-like Growth Factor-I Receptor Monoclonal Antibody) in Combination With CCI-779 (Temsirolimus) in Pediatric Patients With Recurrent or Refractory Solid Tumors
Brief Title: A Phase I Study of IMC-A12 in Combination With Temsirolimus in Pediatric Patients With Recurrent or Refractory Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100175; 10-C-0175
Record Dates: First submitted 2010-08-14; First posted 2010-08-17 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2012-04-04

CONDITIONS: Brain Stem Neoplasms; Glioma; Pinealoma
Keywords: Maximum Tolerated Dose; Dose Escalation; Pharmacokinetics; Antitumor Activity; Biologic Activity
MeSH Terms: conditions — Brain Stem Neoplasms; Glioma; Pinealoma | interventions — cixutumumab; temsirolimus

INTERVENTIONS:
Drug: IMC-A12
Drug: Temsirolimus

SUMMARY:
Background:

- IMC-A12 is an experimental substance designed to inhibit a protein called Type I Insulin-Like Growth Factor Receptor (IGF-1R), which can be found on cancer cells and can promote cancer growth. Temsirolimus is a drug that the U.S. Food and Drug Administration has approved to treat advanced renal cell carcinoma in adults. Researchers do not know if the combination of IMC-A12 and temsirolimus will work in children, but want to determine whether these two drugs may be an effective treatment for recurrent tumors.

Objectives:

* To determine the safety and effectiveness of IMC-A12 and temsirolimus in treating children and adolescents with solid tumors.
* To determine possible side effects of the combination of IMC-A12 and temsirolimus.

Eligibility:

- Children and adolescents between 12 months and 21 years of age who have solid tumors that have not responded to or have relapsed after standard treatment.

Design:

* Participants will be screened with a medical history, physical examination, and imaging studies.
* Participants will receive IMC-A12 and temsirolimus in 28-day cycles of treatment. IMC-A12 will be given as an infusion over 1 hour, once a week, for 4 weeks. Temsirolimus will also be given after IMC-A12 over 30 minutes, once a week, for 4 weeks.
* Participants may continue to receive IMC-A12 and temsirolimus for up to 2 years unless serious side effects develop or the treatment stops being effective.
* Participants will have additional physical exams, blood and urine tests, and imaging studies regularly during each treatment cycle.
* Participants will be followed at regular intervals after the end of the study to collect tumor response and progression data....

DETAILED DESCRIPTION:
Background

* IMC-A12 is a fully recombinant IgG1monoclonal antibody to the insulin-like growth factor receptor (IGFR). It acts as an antagonist of IGF-1 and IGF-2 ligand binding and blocks ligand binding to IGF-1R and inhibits downstream signaling of the two major insulin-like growth factor pathways: MAPK and PI3K/AKT.
* Temsirolimus is a small molecule inhibitor of mTOR, which like rapamycin and everolimus forms a complex with FK506-binding protein (FKBP)12 and mTOR, inhibiting mTOR and leading to anti-proliferative effects, including G1 phase cell cycle arrest and apoptosis.
* Inhibition of mTOR signaling leads to upregulation of IGF-1R signaling which leads to activation of the PI3K/AKT/mTOR pathway. Pediatric pre-clinical models have demonstrated synergistic anti-tumor effects combining IGF-1R antibodies and mTOR inhibitors.

Objectives

* To determine the maximum tolerated dose (MTD) and recommended Phase II dose of IMC-A12 (anti-insulin growth factor-1 receptor monoclonal antibody) administered as an intravenous infusion once weekly in combination with temsirolimus administered intravenously once weekly to children with refractory solid tumors.
* To define the toxicities of the combination regimen and characterize the pharmacokinetics of IMC-A12 in combination with temsirolimus in this patient population.
* Secondary objectives include defining in a preliminary fashion antitumor activity, assessing biologic activity of IMC-A12 and temsirolimus and assessing the incidence of IGFR expression and mTOR pathway activation in recurrent or refractory solid tumors of childhood.

Eligibility

* Patients > 12 months and less than or equal to 21 years of age with a diagnosis and histologic verification (except patients with intrinsic brain stem tumors, optic pathway gliomas or pineal tumors and elevations of serum or CSF alpha-fetoprotein or beta-HCG) of measureable or evaluable relapsed or refractory solid tumors. Current disease state must be one for which there is no known curative therapy, or therapy proven to prolong survival.
* Must have fully recovered from acute toxic effects from all prior therapy, which has been completed within the specified prior time frame.
* Have adequate organ function as determined by laboratory evaluation including normal random or fasting blood glucose within the upper normal limits for age and grade < 2 serum cholesterol and triglyceride levels.
* Subjects with uncontrolled infection, known type I or type II diabetes mellitus, known bone marrow involvement or who have received prior monoclonal antibody therapy targeting IGF-1R or temsirolimus are not eligible.

Design

* This is a phase I study of IMC-A12 administered every 7 days as a 1-hour intravenous infusion at a starting dose of 6 mg/kg. Temsirolimus will be administered intravenously over 30 minutes immediately after IMC-A12 on a once weekly schedule, at a starting dose of 15 mg/m(2).
* One cycle of therapy is considered to be 28 days. Therapy may continue for up to 2 years in the absence of progressive disease or unacceptable toxicity.
* All patients will have required trough blood samples for pharmacokinetic analysis of IMC-A12 and temsirolimus and immunogenicity studies collected at the same time as select routine safety labs. Optional participation in additional pharmacokinetic studies and correlative biology studies will be offered.

ELIGIBILITY:
* Eligibility
* Patients > 12 months and less than or equal to 21 years of age with a diagnosis and histologic verification (except patients with intrinsic brain stem tumors, optic pathway gliomas or pineal tumors and elevations of serum or CSF alpha-fetoprotein or beta-HCG) of measureable or evaluable relapsed or refractory solid tumors. Current disease state must be one for which there is no known curative therapy, or therapy proven to prolong survival.
* Must have fully recovered from acute toxic effects from all prior therapy, which has been completed within the specified prior time frame.
* Have adequate organ function as determined by laboratory evaluation including normal random or fasting blood glucose within the upper normal limits for age and grade < 2 serum cholesterol and triglyceride levels.
* Subjects with uncontrolled infection, known type I or type II diabetes mellitus, known bone marrow involvement or who have received prior monoclonal antibody therapy targeting IGF-1R or temsirolimus are not eligible.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2010-07-28; Primary Completion 2012-04-04 (Actual); Study Completion 2012-04-04 (Estimated)

PRIMARY OUTCOMES:
To determine the MTD and recommended Phase II dose of IMC-A12 (anti-IGFR monoclonal antibody) IV once weekly in combination with temsirolimus IV weekly to children with refractory solid tumors.
To define toxicities and characterize pharmacokinetics.

SECONDARY OUTCOMES:
Define in a preliminary fashion antitumor activity, assess biologic activity of IMC-A12 and temsirolimus and assess the incidence of IGFR expression and mTOR pathway activation in recurrent or refractory solid tumors of childhood.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis D Hickstein, M.D., Principal Investigator — National Cancer Institute (NCI)

REFERENCES:
- [Background] Burtrum D, Zhu Z, Lu D, Anderson DM, Prewett M, Pereira DS, Bassi R, Abdullah R, Hooper AT, Koo H, Jimenez X, Johnson D, Apblett R, Kussie P, Bohlen P, Witte L, Hicklin DJ, Ludwig DL. A fully human monoclonal antibody to the insulin-like growth factor I receptor blocks ligand-dependent signaling and inhibits human tumor growth in vivo. Cancer Res. 2003 Dec 15;63(24):8912-21. PMID 14695208
- [Background] Boulay A, Zumstein-Mecker S, Stephan C, Beuvink I, Zilbermann F, Haller R, Tobler S, Heusser C, O'Reilly T, Stolz B, Marti A, Thomas G, Lane HA. Antitumor efficacy of intermittent treatment schedules with the rapamycin derivative RAD001 correlates with prolonged inactivation of ribosomal protein S6 kinase 1 in peripheral blood mononuclear cells. Cancer Res. 2004 Jan 1;64(1):252-61. doi: 10.1158/0008-5472.can-3554-2. PMID 14729632
- [Background] Majumder PK, Febbo PG, Bikoff R, Berger R, Xue Q, McMahon LM, Manola J, Brugarolas J, McDonnell TJ, Golub TR, Loda M, Lane HA, Sellers WR. mTOR inhibition reverses Akt-dependent prostate intraepithelial neoplasia through regulation of apoptotic and HIF-1-dependent pathways. Nat Med. 2004 Jun;10(6):594-601. doi: 10.1038/nm1052. Epub 2004 May 23. PMID 15156201